CLINICAL TRIAL: NCT02654938
Title: Multicenter, Randomized, Single-blind Safety and Tolerability Clinical Trial of Different Doses of the Immunotherapeutic Drug Mobilan (M-VM3) and Placebo in Patients With Prostate Cancer
Brief Title: Safety and Tolerability Clinical Trial of Different Doses of the Immunotherapeutic Drug Mobilan (M-VM3) and Placebo in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Panacela Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNC-M-VM3-01
Record Dates: First submitted 2015-12-07; First posted 2016-01-13 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; adenovirus; TLR5; immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobilan (M-VM3) (Experimental): Patients with histologically verified non-metastatic prostate cancer (stage 1 or 2) treated with Investigational Drug Product
  Interventions: Drug: Mobilan (M-VM3)
- Placebo (Placebo Comparator): Patients with histologically verified non-metastatic prostate cancer (stage 1 or 2) treated with Placebo (Glucose 5%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mobilan (M-VM3) — Mobilan (M-VM3), innovative experimental drug based on non-replicate adenoviral delivery system consisting genomic vector coding TLR5-receptor and its ligand 502s.
  Arms: Mobilan (M-VM3)
Drug: Placebo — 5% infusion solution of dextrose
  Other Names: Dextrose 5%; Glucose 5%
  Arms: Placebo

SUMMARY:
Phase I single-blinded, randomized, placebo-controlled trial evaluating safety, tolerability, pharmacokinetics and pharmacodynamics of single injections of ascending doses of investigational drug product Mobilan (М-VM3) administered directly into the prostate of patients with prostate cancer.

DETAILED DESCRIPTION:
Mobilan is a type V adenovirus carrying TLR5 receptor and its agonist, protein 502s. It's mechanism of action involves activation of immune system and extensive mobilisation of various immunocytes to administration locus. It's safety and tolerability is currently evaluated in first-in-man phase I study in prostate cancer patients. Treatment strategy for the disease (radical prostatectomy or active observation) will be determined by the Investigator in accordance with routine clinical practice of the hospital.

Patients will be randomised in cohorts of 4 subjects, where 3 subjects will be administered with Mobilan (М-VM3), and one patient will be administered with placebo.

The dose will be escalated from cohort to cohort, the decision on possible dose escalation will be made by Independent Safety Review Board.

ELIGIBILITY:
Inclusion Criteria:

1. Subscribed Informed consent for participation in the trial
2. Men aged 45 to 75 years
3. Patients with histologically verified prostate cancer, stage Т1-Т2, N0, M0
4. Patient's ECOG status 0-2
5. Negative tests for serologic markers of HIV-infection, viral hepatitis В and С, syphilis Patient and his partner should agree to use barrier contraception throughout the study period

Exclusion Criteria:

1. Failure to obtain Informed consent
2. Clinical or radiological signs of metastases
3. Indication to hormone therapy of prostate cancer
4. Clinically significant cardiovascular diseases:

   * Myocardial infarction within 6 months prior the screening
   * Unstable stenocardia within 3 months prior the screening
   * Severe circulation failure (FC III)
   * Clinically significant arrhythmias
   * Hypotension (systolic blood pressure < 86 mm Hg) or bradycardia with HR < 50 beats per min.
   * Uncontrolled arterial hypertension (systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg.)
5. Clinically significant CNS diseases at the screening
6. Current infection or another severe or systemic disease which increases risk of treatment sequelae
7. Pituitary gland or adrenal disorders in medical history
8. Other malignant tumors within the last 5 years
9. Other concomitant diseases in medical history which according to Investigator may aggravate during the study, including uncontrolled diabetes mellitus, rectal diseases, rectal fissures, hemorrhoid, rectal polyps, rectostenosis, inflammatory urinary diseases: chronic prostatitis, cystitis, urethral catheter, chronic urine retention.
10. Complicated allergic history, systemic allergic reaction, any dietary allergy, intolerability, limitations or specific diets which according to the Investigator may be a contraindication for subject participation in the present study.
11. Administration of drug products which have a marked effect on immune system within 3 previous months prior the screening, long-term intake of disaggregants (warfarin, low molecular heparin except for ThromboASS).
12. Participation in other clinical studies or administration of investigational drug products within 30 days prior the screening, or persisting adverse reactions of any investigational drug product.
13. Any clinically significant patient's health disorders and/or laboratory abnormalities not enlisted in the Protocol which are identified at the screening, and/or any reason which according to the Investigator may prevent the patient's participation in the study.
14. Drug or alcohol abuse at the screening or in the past which according to the Investigator makes the patient ineligible for participation in the study: intake of more than 5 units of alcohol a week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of vine or 50 ml of alcohol) or anamnestic data on alcoholism, narcomania, drug abuse and/or history of significant alcohol or drug abuse inducing drug dependence, within one year prior the screening visit.
15. Vaccination made 14 days prior the study
16. Smoking of more than 10 cigarettes a day
17. Unability to understand or follow study instructions
18. Lack of availability during 29 days after administration of the investigational drug product, fails to follow visit schedule
19. Individual intolerability of the investigational drug product components

Study withdrawal criteria:

1. Any patient may refuse from the study participation on his own wish in any moment on any study stage.
2. Principal Investigator may withdraw any patient from the study in the following cases:

   * Investigator makes the decision that a patient should be withdrawn in his own best interests
   * Patient develops any serious adverse reactions/events in the screening period
   * Patient has been enrolled to the study with violations, or does not follow the protocol requirements
   * Patient needs additional treatment in the screening period
3. Sponsor has right to terminate the study in any moment.
4. Regulatory authorities have right to terminate the study in any moment.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of adverse events (according to CTCAE v 4.03 classification) | Baseline to up to 29 days after the drug administration

SECONDARY OUTCOMES:
Exposure of Mobilan DNA vector in patient's peripheral blood | Baseline to up to 29 days after the drug administration
  Using validated PCR assay
Prostate-specific antigen (PSA) measure | On Day 29 after the drug administration
  Baseline PSA level will be taken from medical history
Immune cell count in whole blood of patients assessed with flow cytometry | Baseline to up to 29 days after the drug administration
  Including leucocytes, lymphocytes, T-lymphocyte, leukocyte index, total T-lymphocytes, CD3, T-helper cells CD3 + CD4 +, T-cytotoxic CD3 + CD8 +, regulation index (CD4 / CD8), double-cells CD4 + / CD8 +, NK cells CD3-CD (16 + 56) +, TNK-cells CD3 + CD (16 +56) +, B-lymphocytes CD19 +, 0-lymphocytes
Histopathological assessment of prostate tissue using Gleason grading system (if prostatectomy is made in the study period, and material is available for analysis) | On Day 29 after the drug administration
  The Gleason grading system is used to evaluate the stage of prostate cancer using samples from biopsy or post-surgical samples as follow:
  1 - The cancerous prostate closely resembles normal prostate tissue. 2 - The tissue still has well-formed glands, but they are larger and have more tissue between them. 3 - The tissue still has recognizable glands, but the cells are darker. 4 - The tissue has few recognizable glands. 5 - The tissue does not have any or only a few recognizable glands.
Presence of protein 502s in blood plasma | Baseline to up to 29 days after the drug administration
  Using ELISA assay
Titer of 502 antibodies (AB) in peripheral blood serum | Baseline to up to 29 days after the drug administration
  Using ELISA assay
Histopathological assessment of prostate tissue using Irani scale (if prostatectomy is made in the study period, and material is available for analysis) | On Day 29 after the drug administration
  Irani J (1997) scale include histological assessment of slide mounts obtained after operation as follow:
  Degree of immune cell infiltration:
  0 - No inflammatory cells, 1 - Scattered inflammatory cell infiltrate within the stroma without lymphoid nodules, 2 - Nonconfluent lymphoid nodules, 3 - Large inflammatory areas with confluence of infiltrate

CONTACTS AND LOCATIONS:
Overall Officials: Vsevolod B. Matveev, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Russian Oncological Research Center named after N. N. Blokhin" of the Russian Academy of Medical Sciences; Boris Y. Alexeev, MD, PhD, Principal Investigator — Moscow Scientific Research Institute of Oncology named after P. A. Hertsen of the Ministry of Health of the Russian Federation; Vladimir M. Moiseenko, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Saint Petersburg Clinical Scientific and Practical Center for Special types of medical care (Oncological)"; Sergey V. Mishugin, MD, PhD, Principal Investigator — Moscow State Budgetary Healthcare Institution "City Clinical Hospital № 57" of Moscow Healthcare Department; Alexander K. Nosov, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Scientific Research Oncology Institute named after N.N. Petrov" of the Ministry of Health of the Russian Federation; Dmitry Y. Pushkar, MD, PhD, Principal Investigator — Moscow State University of Medicine and Dentistry
Locations (6):
- Russia (6):
  - Federal State Budgetary Institution "Russian Oncological Research Center named after N. N. Blokhin" of the Russian Academy of Sciences, Moscow
  - Moscow Scientific Research Institute of Oncology named after P. A. Hertsen of the Ministry of Health of the Russian Federation, Moscow
  - Moscow State Budgetary Healthcare Institution "City Clinical Hospital № 57" of Moscow Healthcare Department, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - Federal State Budgetary Institution "Saint Petersburg Clinical Scientific and Practical Center for Special types of medical care (Oncological)", Saint Petersburg
  - Federal State Budgetary Institution "Scientific Research Oncology Institute named after N.N. Petrov" of the Ministry of Health of the Russian Federation, Saint Petersburg